CLINICAL TRIAL: NCT05154890
Title: A Phase 1/2 Multiple Ascending-Dose Study in Subjects With Homocystinuria Due to Cystathionine β-Synthase (CBS) Deficiency to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of ACN00177
Brief Title: A Multiple Ascending Dose Study of ACN00177 (Pegtarviliase) in Subjects With CBS Deficiency
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Aeglea Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CACN00177-100D; 2019-004791-19 (EudraCT Number)
Record Dates: First submitted 2021-08-20; First posted 2021-12-13 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Homocystinuria Due to Cystathionine Beta-Synthase Deficiency
MeSH Terms: conditions — Homocystinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Pegtarviliase Cohort 1 (Experimental): Planned for 4 subjects ≥18 years of age dosing at Dose A weekly for a total of 4 doses
  Interventions: Drug: Pegtarviliase IV
- Pegtarviliase Cohort 2 (Experimental): Planned for 4 subjects ≥12 years of age dosing at Dose B weekly for a total of 4 doses
  Interventions: Drug: Pegtarviliase SC
- Pegtarviliase Cohort 3 (Experimental): Planned for 4 subjects ≥12 years of age (≥18 in the US) dosing at Dose C weekly for a total of 4 doses
  Interventions: Drug: Pegtarviliase SC
- Pegtarviliase Cohort 4 (Experimental): Planned for 4 subjects ≥12 years of age (≥18 in the US) dosing at Dose D weekly for a total of 4 doses
  Interventions: Drug: Pegtarviliase SC
- Pegtarviliase Cohort 5 (Experimental): Optional cohort for up to 12 subjects ≥12 years of age (≥18 in the US) dosing at Dose E weekly for a total of 13 doses
  Interventions: Drug: Pegtarviliase SC

INTERVENTIONS:
Drug: Pegtarviliase IV — Administered IV
  Other Names: ACN00177
  Arms: Pegtarviliase Cohort 1
Drug: Pegtarviliase SC — Administered SC
  Other Names: ACN00177
  Arms: Pegtarviliase Cohort 2; Pegtarviliase Cohort 3; Pegtarviliase Cohort 4; Pegtarviliase Cohort 5

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of pegtarviliase in approximately 36 subjects with homocystinuria due to CBS deficiency.

DETAILED DESCRIPTION:
The purpose of this Phase 1/2 study is to evaluate the safety, pharmacokinetics and pharmacodynamics of multiple ascending doses of pegtarviliase in subjects with homocystinuria due to CBS deficiency. The study is composed of 2 parts: Part 1: a single IV (intravenous) cohort with 4 once-weekly (QW) doses of study drug and Part 2: three SC (subcutaneous) cohorts with 4 QW doses of study drug, with an optional fifth.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of homocystinuria due to CBS deficiency
2. Capable of providing signed informed consent/assent and to comply with all study related procedures
3. Is ≥12 years of age (≥18 in the US) at the time of signing the informed consent/assent
4. Plasma tHcy ≥50 µM (rounded to the nearest whole number) and documentation of previous tHcy ≥80 µM
5. Female subjects of child-bearing potential must have a negative serum pregnancy test during the screening period and a negative urine pregnancy test prior to dosing on the first day of treatment
6. If the subject (male or female) is engaging in sexual activity, he/she must be unable to become pregnant/cause pregnancy or must agree to use highly effective contraception
7. Subjects receiving pyridoxine and/or betaine must be on the same dose of the medication(s) for at least 6 weeks prior to the first administration of study drug and be willing and able to remain on a stable dose for the duration of the study. Similarly, those on prescribed dietary therapy must be on a consistent dietary regimen for at least 6 weeks prior to study drug and should maintain this regimen for the duration of the study

Exclusion Criteria:

1. Other medical conditions or co-morbidity(ies) that, in the opinion of the investigator, would put the subject at increased medical risk or interfere with study compliance or data interpretation (eg, severe intellectual disability that precludes completion of the required study assessments)
2. Currently participating in another therapeutic clinical study or has received any investigational agent within 30 days or 5 half-lives, whichever is longer, prior to the first dose of study drug in this study
3. Surgery requiring general anesthesia within 8 weeks prior to the first dose of study drug or planned surgery druing the treatment period
4. Active infection requiring anti-infective therapy <2 weeks prior to the first dose of study drug in this study; anti-infective therapy that completes ≥2 weeks prior to first dose of study drug is acceptable
5. Pregnant or nursing
6. Females of child-bearing potential who are using or plan to use estrogen-containing contraception during the study (unless the subject currently using estrogen-containing contraceptives is willing to switch to a non-estrogen-containing contraceptive at least 1 week before dosing and for the duration of the study) and for 30 days after the last dose
7. History of hypersensitivity to polyethylene glycol (PEG) that, in the judgment of the investigator, puts the subject at unacceptable risk for adverse events (AEs)
8. Serum creatinine level >1.5× the upper limit of normal (ULN)
9. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin level > 2× the ULN

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Reporting will be from signing consent through study completion, an average of 70 days
  Incidence of treatment-emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetic Profile of IV pegtarviliase Cmax | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  Cmax
Pharmacokinetic Profile of IV pegtarviliase AUC | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  AUC
Pharmacokinetic Profile of IV pegtarviliase Tmax | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  Tmax
Pharmacokinetic Profile of IV pegtarviliase T1/2 | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  T1/2
Pharmacokinetic Profile of Subcutaneous pegtarviliase Cmax | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  Cmax
Pharmacokinetic Profile of Subcutaneous pegtarviliase AUC | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  AUC
Pharmacokinetic Profile of Subcutaneous pegtarviliase Tmax | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  Tmax
Pharmacokinetic Profile of Subcutaneous pegtarviliase T 1/2 | At pre-dose, 1hour, 6hours, 24hours, 48hours, 72hours, 96hours and 120hours
  T1/2
Changes in total plasma homocysteine after treatment with pegtarviliase | At Visit Day 29
  Changes in total plasma homocysteine after treatment with pegtarviliase
Time course of tHcy change after pegtarviliase administration and reversibility upon follow up post dosing | Weekly, baseline through study completion, up to 12 weeks
  Time course of tHcy change after pegtarviliase administration and reversibility upon follow up post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Cortney Caudill, Study Director — Aeglea Biotherapeutics
Locations (9):
- UT Southwestern Medical Center, Dallas, Texas, United States
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- United Kingdom (5):
  - University Hospitals Birmingham NHS, Birmingham
  - Great Ormond Street Hospital, London
  - Guy's and St Thomas' Hospital NHS Foundation Trust, London
  - University College London, London
  - Salford Royal NHS Foundation Trust, Salford